CLINICAL TRIAL: NCT00491582
Title: The Effect of Growth Hormone (GH) on Intramyocellular Lipids (IMCL), Intrahepatocellular Lipids (IHCL) and Visceral Fat Mass in Relation to Insulin Resistance
Brief Title: The Effects of Growth Hormone (GH) on Lipid Depots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Emanuel Christ, Prof. Emanuel Christ, MD, PhD, Insel Gruppe AG, University Hospital Bern
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 320000-109522/1
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Athletes, controls, patients (No Intervention): Sedentary controls: age, BMI, Gender and waist matched (to the growth hormone deficient patients) healthy control subjects Endurance trained athletes: minimal >50 mlO2/KG body weight
  Interventions: Drug: Growth hormone replacement therapy in growth hormone deficient patients only.

INTERVENTIONS:
Drug: Growth hormone replacement therapy in growth hormone deficient patients only. — Genotropin once/daily sc., titration scheme according to the consensus guidelines of the GH and IGF-research society Duration: 6 months
  Other Names: Genotropin

SUMMARY:
This study aims at investigating the effect of growth hormone on lipid-content of muscle and liver as well as visceral fat mass in relation to insulin sensitivity.

In addition, hormonal regulation and free fatty availability is assessed during a physical exercise at 50-60% VO2max.

Finally, the value of physical exercise in diagnosing growth hormone deficiency is investigated.

Hypothesis: 1) Lipid content of muscle and liver change with physical exercise and exercise capacity and free fatty availability will influence these changes. 2)Growth hormone replacement therapy will predominantly reduce visceral fat mass and increase free fatty availability.

3)Free fatty availability during exercise will be reduced in growth hormone deficient patients 4)Physical exercise may be an alternative way to diagnose growth hormone deficiency

DETAILED DESCRIPTION:
Using the two-step hyperinsulinaemic-euglycaemic clamp technique hepatic and peripheral insulin sensitivity is assessed.

Lipid depots (skeletal muscle and liver) are measured by MR-spectroscopy, visceral fat mass by MR-imaging.

Exercise capacity ist measured on a treadmill. Counterregulatory hormones, glucose and free fatty acids are measured during a 2h physical exercise at 50-60 VO2max Identical investigations are performed in adult growth hormone (GH) deficient patients before and after six months GH replacement therapy, in sedentary matched control subjects and in endurance trained athletes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with proven GH-deficiency defined as a peak GH of less than 3mU/l during an insulin provocation test with nadir plasma glucose less than 2.2 mmol/l and additionally, stable conventional replacement therapy including corticoids, thyroxin and gonadal hormones as needed.
* Ability to perform an exercise test on a treadmill or a walking band.
* Willingness to participate in the study and to give written informed consent.

Exclusion Criteria:

Active neoplasia

* Severe cardiovascular disease (unstable coronary heart disease, heart failure NYHA III-IV)
* Type 2 Diabetes mellitus
* Haemophilia or other coagulation disorder
* Inability to exercise
* Contraindications to exposure to a 3-T magnetic field (Pace-Makers, osteosynthetic material)
* Pregnant women
* Women in childbearing age unless on a continuous contraceptive therapy or surgically sterilised.
* Abnormal liver or renal function (Creatinine >130mmol/L, normal reference 45-93mmol/L; ASAT and ALAT > 3 times the upper reference limit).
* Major depression, psychosis and other severe personality disorders
* Excessive alcohol consumption (>60g/d) or drug-abuse
* Refusal to give written consent
* Patients, who are not suitable for the study according to the study physician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Determination of visceral fat mass by MRI,Determination of IMCL and IHCL by MR Spectroscopy, Determination of peripheral and hepatic insulin sensitivity by two step hyperinsulinemic euglycemic clamp | 2008 - 2009

SECONDARY OUTCOMES:
maximal exercise capacity | 2008 - 2009
Measurement of serum alphaKlothe by an ELISA | 2008 - 2013
  Measured in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel R Christ, Prof,MD,PhD, Principal Investigator — Abt. für Endokrinologie, Diabetologie und Klin. Ernährung, Inselspital, Berne
Locations (1):
- Abt. für Endokrinologie, Diabetologie und Klin. Ernährung, Inselspital, Bern, Switzerland

REFERENCES:
- [Derived] Egger A, Kreis R, Allemann S, Stettler C, Diem P, Buehler T, Boesch C, Christ ER. The effect of aerobic exercise on intrahepatocellular and intramyocellular lipids in healthy subjects. PLoS One. 2013 Aug 14;8(8):e70865. doi: 10.1371/journal.pone.0070865. eCollection 2013. PMID 23967125